CLINICAL TRIAL: NCT07107022
Title: i-RISE: International Acute Ischemic Stroke Study With the Penumbra System®
Brief Title: Study to Collect Real-world Performance and Safety Data on Penumbra System® in Population With Acute Ischemic Stroke (AIS).
Acronym: i-RISE
Status: Recruiting | Type: Observational
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP 30324
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke (AIS)
Keywords: Penumbra System; Thrombectomy; Penumbra ENGINE®; mechanical thrombectomy; Neuro Thrombectomy; Neurovascular Catheters
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients with acute ischemic stroke (AIS): Device: Penumbra System®
  Interventions: Device: Penumbra System ®

INTERVENTIONS:
Device: Penumbra System ® — Neurovacular Mechanical Thrombectomy with the Penumbra System®

SUMMARY:
The primary objective of this study is to collect real-world performance and safety data on the Penumbra System in a patient population with acute ischemic stroke (AIS)

DETAILED DESCRIPTION:
Post-market, real-world, prospective, single-arm, multi-center study that will enroll up to 200 participants at up to 15 sites globally

ELIGIBILITY:
Inclusion Criteria:

* I.1. Patient age 18-75 years
* I.2. Pre-stroke mRS 0-1
* I.3. Patients experiencing acute ischemic stroke who are eligible for mechanical thrombectomy using the Penumbra System
* I.4. Frontline treatment with Penumbra System
* I.5. Signed informed consent per Institution Review Board/Ethics Committee

Exclusion Criteria:

* E.1. Alberta Stroke Program Early CT Score (ASPECTS) ≤6 (for anterior circulation strokes)
* E.2. Any comorbid disease or condition expected to compromise survival or ability to complete follow-up assessments through 90 days
* E.3. Currently participating in an investigational (drug, device, etc.) clinical trial that will influence the endovascular procedure or acute treatment of the patient. Patients in secondary prevention, observational, natural history, and/or
* epidemiological studies are eligible.
* E.4. Other medical, behavioral, or psychological conditions that in the opinion of the Investigator could limit the patient's ability to participate in the study, including compliance with follow-up requirements, or that could impact the scientific integrity of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with acute ischemic stroke (AIS) who are eligible for aspiration based mechanical thrombectomy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Outcomes: | It is anticipated this study will take approximately 2 years. All participants will be followed for approximately 90-day or to outcome (e.g., withdrawal, death), whichever occurs first.
  Angiographic revascularization of the occluded target vessel immediately post- procedure as defined by modified Thrombolysis in Cerebral Infarction (mTICI) 2b or higher Angiographic revascularization of the occluded target vessel immediately post- procedure as defined by mTICI 2c or higher
  * Angiographic revascularization of the occluded target vessel after the first pass as defined by mTICI 2b or higher
  * Angiographic revascularization of the occluded target vessel after the first pass as defined by mTICI 2c or higher

CONTACTS AND LOCATIONS:
Overall Officials: Marios Nikos Psychogios, MD, Principal Investigator — University Hospital of Basel, Switzerland
Locations (2):
- Sir Charles Gairdner Hospital, Nedlands, Western Australia, Australia
- Universitätsspital Basel, Basel, Basel-Landschaft, Switzerland

IPD SHARING:
Plan to Share IPD: No